CLINICAL TRIAL: NCT04856436
Title: Maternal and Neonatal Outcomes Following Benzodiazepine Use During Pregnancy
Brief Title: Maternal and Neonatal Outcomes Following Exposure to Benzodiazepines During Pregnancy
Status: Completed | Type: Observational
Sponsor: Sungkyunkwan University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Ju-Young Shin, Associate Professor, Sungkyunkwan University
Other Study IDs: SKKU-2021-PREG-BZ
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Related; Benzodiazepines Causing Adverse Effects in Therapeutic Use; Congenital Anomaly
MeSH Terms: conditions — Congenital Abnormalities | interventions — Benzodiazepines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with exposure to benzodiazepines: Women who gave birth during 2011-2018, were aged 20-45 years and were filled at least one benzodiazepine prescription during the first trimester (first 90 days of pregnancy).
  Interventions: Drug: Benzodiazepine
- Pregnant women without exposure to benzodiazepines: Women who gave birth during 2011-2018, were aged 20-45 years and did not fill a benzodiazepine prescription during the 3 months before the pregnancy onset through the end of the first trimester
  Interventions: Drug: Benzodiazepine

INTERVENTIONS:
Drug: Benzodiazepine — Exposure to benzodiazepine during early pregnancy

SUMMARY:
This is a nationwide cohort study to assess maternal and neonatal outcomes following exposure to benzodiazepines during pregnancy.

DETAILED DESCRIPTION:
Benzodiazepines are widely used in pregnant women; however, their safety on congenital malformations in a real-world setting is still uncertain. We aimed to assess the association between benzodiazepine use in early pregnancy and the risk of congenital malformations. We will conduct a retrospective nationwide cohort study using the Health Insurance Review and Assessment (HIRA) database of South Korea, which covers the entire South Korean population.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancies with live birth, 2011-2018
* Pregnancies linked to liveborn infants
* Pregnancies aged 20-45 years at delivery

Exclusion Criteria:

* Pregnancies with a chromosomal abnormality
* Pregnancies with exposure to known teratogenic drugs (e.g. antineoplastic agent, warfarin, lithium, isotretinoin, misoprostol, thalidomide) during the first trimester
* Pregnancies with no benzodiazepine prescription during the first trimester, but with at least one benzodiazepine prescription during the 3 months before the pregnancy onset

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who gave birth in South Korea between 2011 and 2018
Sampling Method: Probability Sample
Enrollment: 3094227 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Risk of congenital malformations | from the birth date until up to 8 years, death, or study end date (Dec 31, 2019)
  Overall congenital malformations and organ-specific congenital malformations in infants, which are confirmed by diagnostic records in the HIRA database. All infants were followed up for at least 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Young Shin, PhD, Principal Investigator — Sungkyunkwan University
Locations (1):
- Sungkyunkwan University, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellantuono C, Tofani S, Di Sciascio G, Santone G. Benzodiazepine exposure in pregnancy and risk of major malformations: a critical overview. Gen Hosp Psychiatry. 2013 Jan-Feb;35(1):3-8. doi: 10.1016/j.genhosppsych.2012.09.003. Epub 2012 Oct 6. PMID 23044244
- [Background] Grigoriadis S, Graves L, Peer M, Mamisashvili L, Dennis CL, Vigod SN, Steiner M, Brown C, Cheung A, Dawson H, Rector N, Guenette M, Richter M. Benzodiazepine Use During Pregnancy Alone or in Combination With an Antidepressant and Congenital Malformations: Systematic Review and Meta-Analysis. J Clin Psychiatry. 2019 Jul 9;80(4):18r12412. doi: 10.4088/JCP.18r12412. PMID 31294935
- [Background] Bais B, Molenaar NM, Bijma HH, Hoogendijk WJG, Mulder CL, Luik AI, Lambregtse-van den Berg MP, Kamperman AM. Prevalence of benzodiazepines and benzodiazepine-related drugs exposure before, during and after pregnancy: A systematic review and meta-analysis. J Affect Disord. 2020 May 15;269:18-27. doi: 10.1016/j.jad.2020.03.014. Epub 2020 Mar 5. PMID 32217339
- [Background] Iqbal MM, Sobhan T, Ryals T. Effects of commonly used benzodiazepines on the fetus, the neonate, and the nursing infant. Psychiatr Serv. 2002 Jan;53(1):39-49. doi: 10.1176/appi.ps.53.1.39. PMID 11773648
- [Background] Shyken JM, Babbar S, Babbar S, Forinash A. Benzodiazepines in Pregnancy. Clin Obstet Gynecol. 2019 Mar;62(1):156-167. doi: 10.1097/GRF.0000000000000417. PMID 30628916
- [Derived] Noh Y, Lee H, Choi A, Kwon JS, Choe SA, Chae J, Kim DS, Shin JY. First-trimester exposure to benzodiazepines and risk of congenital malformations in offspring: A population-based cohort study in South Korea. PLoS Med. 2022 Mar 2;19(3):e1003945. doi: 10.1371/journal.pmed.1003945. eCollection 2022 Mar. PMID 35235572